CLINICAL TRIAL: NCT05304000
Title: Psychophysiological Effects of Controlled Respiration: Noninvasive Relaxation Techniques
Brief Title: Psychophysiological Effects of Controlled Respiration and Mindfulness
Acronym: PECRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Spiegel, Professor, Department of Psychiatry and Behavioral Sciences, Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41398
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Stress, Physiological; Stress, Emotional; Insomnia
Keywords: stress; breathwork; mindfulness meditation; mood; anxiety; wearable; physiology
MeSH Terms: conditions — Stress, Psychological; Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Randomized prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness Meditation (Active Comparator): 5 minutes a day of mindfulness meditation practice for 28 days (passive attention to breath) delivered remotely through a video link.
  Interventions: Behavioral: Mindfulness Meditation
- Cyclic Sighing Breathing (Experimental): 5 minutes a day of active breathwork practice for 28 days delivered remotely through a video link. The protocol consists of slow inhales until lungs felt full then one more inhale to maximally fill the lungs, followed up a slow exhale. Repeat this cycle for 5 minutes.
  Interventions: Behavioral: Cyclic Sighing Breathing
- Box Breathing (Experimental): 5 minutes a day of active breathwork practice for 28 days delivered remotely through a video link. The protocol consists of equal duration of inhale, hold, exhale, hold cycles. The duration of the cycle is determined by the participant's comfort level with holding. (e.g. 4 sec inhale, 4 sec hold, 4 sec exhale, 4 sec hold). Repeat this cycle for 5 minutes.
  Interventions: Behavioral: Box Breathing
- Cyclic Hyperventilation with Retention (Experimental): 5 minutes a day of active breathwork practice for 28 days delivered remotely through a video link. The protocol consists of 30 breaths (inhale deeply through the nose and exhale passively through the mouth) and after those 30 breaths, to exhale all their air via their mouth and to calmly wait with lungs empty for 15 seconds. Repeat this cycle for 5 minutes.
  Interventions: Behavioral: Cyclic Hyperventilation with Retention

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Participants are informed they should sit down in a chair or, if they preferred, to lie down, and then to set a timer for 5 minutes. Then they are told to close their eyes and to start breathing while focusing their mental attention on their forehead region between their two eyes. They are told that if their focus drifted from that location to re-recenter their attention by focusing back first on their breath and then on the forehead region between their eyes. They are told that as thoughts arise, to recognize that as normal, refocus their attention back to their forehead region and to continue the practice until time has elapsed.
  Arms: Mindfulness Meditation
Behavioral: Cyclic Sighing Breathing — Participants are informed they should sit down in a chair or, if they prefer, to lie down, and to set a timer for 5 minutes. Then they are told to inhale slowly, and that once their lungs are expanded, to inhale again once more to maximally fill their lungs -- even if the second inhale was shorter in duration and smaller in volume than the first, and then to slowly and fully exhale all their breath. They are told to repeat this pattern of breathing for 5 minutes. They are also informed that ideally, both inhales would be performed via their nose and the exhale would be performed via their mouth, but that if they preferred, they are welcome to do the breathing entirely through their nose. They are also informed that it is normal for the second inhale to be briefer than the first.
  Arms: Cyclic Sighing Breathing
Behavioral: Box Breathing — Participants are informed they should sit down in a chair or lie down, and to get a timer. Then they are told to take the "CO2 tolerance test" as follows: Take 4 breaths through the nose. Then take a maximally deep breath and once your lungs are full, exhale as slowly as possible through your nose or mouth. Time how long it takes to empty your lungs; this will be your C02 discard duration. Use your discard duration to determine how long your inhales, exhales, and breath holds should be (CO2 discard time) by using this table: <20 sec = 3 - 4 sec, 25 - 45 sec = 5 - 6 sec, 50 - 75+ sec = 8 -10 sec. They are then told to inhale, hold, exhale, hold (for the duration determined by the C02 discard table) and to repeat this pattern for the entire 5 minutes. If at any point they had to strain to reach these times, they should simply reduce the duration of inhales, exhales, and breath holds. We ask participants to perform all breathing through their nose, if possible.
  Arms: Box Breathing
Behavioral: Cyclic Hyperventilation with Retention — Participants are informed they should sit down in a chair or, if they prefer, to lie down, and to set a timer for 5 min. Then they are told to inhale deeply (ideally through their nose but if that is not possible, to inhale through their mouth) and then exhale by passively letting the air "fall out from the mouth". We inform them that for sake of this protocol, that pattern of a deep inhale through the nose and passively letting the air "fall out from the mouth" = 1 breath.
  Then they are instructed to perform 30 breaths (in and out) in this manner, and after those 30 breaths, to exhale all their air via their mouth and to calmly wait with lungs empty for 15 seconds.
  Arms: Cyclic Hyperventilation with Retention

SUMMARY:
The investigators aim to understand the effectiveness of 3 types of breathwork exercises and a mindfulness meditation control on improving psychological and physiological measures of wellbeing. The interventions will be delivered remotely and effects are monitored through daily surveys and physiological monitoring with WHOOP wristband through a 28-day period. The information gained will help develop the most effective remote interventions for lowering stress and improving wellbeing. The study will be run on a healthy general population. The three breathing conditions were 1) Cyclic Sighing, which emphasizes relatively prolonged exhalations, 2) Box Breathing, which is equal duration of inhalations, breath retentions, exhalations and breath retentions, and 3) Cyclic Hyperventilation with Retention, with longer, more intense inhalations and shorter, passive exhalations. Mindfulness Meditation practice involved passive attention to breath.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine psychological and physiological effects of breathwork in general in comparison to mindfulness meditation.

SECONDARY OBJECTIVES:

I. Examine the effectiveness of specific breathwork protocols in improving mood and physiological wellness metrics in comparison to mindfulness meditation.

OUTLINE:

Of 140 potential participants who consented, 134 were randomized to the four interventions (3 were lost to follow-up and 3 were excluded due to lack of WHOOP straps at this stage). Out of the 134 that were randomized, 108 were enrolled. The primary reasons for attrition at this stage were due to pandemic-related reasons or loss of contact with the participants.

From the 108 subjects enrolled, 24 were randomized into the Mindfulness Meditation control condition and 84 were randomized to the treatment conditions (30 Cyclic Sighing, 21 Box Breathing, 33 Cyclic Hyperventilation with Retention). The initial randomization consisted of a permuted block randomization design with a block size of eight.

Both prior to and after the 28-day intervention, participants completed two brief questionnaires to assess the impact of the intervention on the daytime sequelae of sleep and anxiety: PROMIS Sleep Related Impairment - Short Form 8a, and the State-Trait Anxiety Questionnaire. Participants also completed a debriefing questionnaire at the end of the study. During the 28-day intervention period, participants did their assigned 5-minute exercise and completed two questionnaires before and after, the State Anxiety Inventory and the Positive and Negative Affect Schedule (PANAS). Participants received invitations to instructional videos (pre-recorded by Andrew D. Huberman) on the breathing exercises 3-5 days prior to the start of the study as well as daily text messages that reminded them to complete their exercises and pre-and-post-practice assessments. They were asked to complete the exercises only once a day.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Not pregnant
* Able to follow basic instruction for prescreen and scheduling
* Compliant with investigator instructions during the consent process and participation in the study

Exclusion Criteria:

* Age <18
* Pregnant
* Non-English speaking
* Anyone with personality disorders or psychosis such as schizoaffective disorder
* Demonstrates evidence of severe psychiatric disorder in prescreen or email contact (as judged by Dr. Spiegel)
* Glaucoma
* History of seizures
* Suicidal
* Heart disease (based on PI's clinical judgement, dependent on the severity of the symptoms)
* Current untreated psychosis, or bipolar disorder, or substance/alcohol abuse/dependence (based on PI's clinical judgement, dependent on the severity of the symptoms)
* Any Medical condition that could be exasperated by study participation (based on PI's clinical judgement)
* Non USA mailing address to receive the WHOOP strap
* Vision or hearing impairment severe enough to interfere with study participation,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
State Anxiety | Daily from Day 0 to 29
  STAI State Trait Anxiety
Trait Anxiety | Day 0 and Day 29 (Baseline and Endpoint)
  STAI State Trait Anxiety
Positive Affect | Daily from Day 1 to 28
  PANAS Positive Affect
Negative Affect | Daily from Day 1 to 28
  PANAS Negative Affect
Daytime Sleep Related Disturbance | Day 0 and Day 29 (Baseline and Endpoint)
  PROMIS Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 8a PROMIS Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 8a PROMIS Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 8a PROMIS Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 8a PROMIS Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 8a PROMIS Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 8a PROMIS Sleep Related Impairment Short Form 8a
Resting Heart Rate | Daily from Day 1 to 28
  Daily obtained from WHOOP wrist band
Heart Rate Variability | Daily from Day 1 to 28
  Daily obtained from WHOOP wrist band
Respiratory Rate | Daily from Day 1 to 28
  Daily obtained from WHOOP wrist band
Sleep Duration | Daily from Day 1 to 28
  Daily obtained from WHOOP wrist band
Change in number of hours of sleep | Daily from Day 1 to 28
  Daily obtained from WHOOP wrist band as Hours of Sleep. Changes in the hours of sleep will be assessed with more hours indicating better sleep.
Change in the ratio of number of hours of sleep to hours in bed | Daily from Day 1 to 28
  Obtained daily from WHOOP wrist band as sleep efficiency. Changes in the Whoop Sleep Efficiency score will be assessed with higher score (ratio) indicating higher sleep efficiency.

SECONDARY OUTCOMES:
Adherence to Protocol | Daily from Day 1 to 28
  Number of days subjects did their exercises out of the 28 days assigned

OTHER OUTCOMES:
Debriefing survey | Day 29 (study endpoint)
  Open ended survey about how subjects would describe the protocols

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, M.D., Principal Investigator — Professor of Psychiatry, Stanford University; Andrew Huberman, Ph.D., Principal Investigator — Stanford University; Manuela Kogon, M.D., Study Director — Stanford University
Locations (2):
- United States (2):
  - Neurobiology and Ophthalmology, Palo Alto, California
  - Dept. of Psychiatry, Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT05304000/SAP_000.pdf
  • Informed Consent Form (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT05304000/ICF_001.pdf